CLINICAL TRIAL: NCT06042296
Title: Expression of CD44, PCNA and E-cadherin in Pterygium Tissue
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, HUMEYRA YILDIRIM, Expression of CD44, PCNA and E-cadherin in pterygium tissue, Balikesir University
Other Study IDs: BAUNHYILDIRIM-1
Record Dates: First submitted 2023-09-10; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Pterygium
Keywords: PCNA,; cd44; e-cadherin; immunohistochemistry; pterygium
MeSH Terms: conditions — Pterygium | interventions — Cadherins; Proliferating Cell Nuclear Antigen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control group: group 1 -control group normal conjunctiva from 30 patients
  Interventions: Other: Expression of CD44, E-cadherin and PCNA
- group 2 primary pterygia: primary pterygia samples from 30 patients
  Interventions: Other: Expression of CD44, E-cadherin and PCNA
- group 3 recurrent pterygia: recurrent pterygia samples from 30 patients
  Interventions: Other: Expression of CD44, E-cadherin and PCNA

INTERVENTIONS:
Other: Expression of CD44, E-cadherin and PCNA — The investigators use primary antibodies against CD44 (1:50 dilution) and E-cadherin (1:200 dilution), and a human monoclonal antibody against PCNA (1:100 dilution) for antigen retrieval. Histopathological and immunohistochemical staining findings will be reported using a Nikon light microscope and an image analysis system (Nikon Instruments Europe BV)

SUMMARY:
Purpose: Pterygium is a common ocular surface disease defined by fibrovascular conjunctival growth extending onto the cornea. Its pathogenesis remains unclear. In severe cases, it may extend into the central cornea, inducing irregular corneal astigmatism and causing loss of vision. CD44( phagocytic glycoprotein-1 ) is involved in the organization of certain cellular processes, for instance, cell adhesion, division, and migration, by binding with its main ligand, hyaluronic acid. Proliferating cell nuclear antigen (PCNA) is a proliferation marker in the nucleus. E-cadherin is a calcium-dependent transmembrane glycoprotein that plays a significant role in the protection of tissue integrity and cell-to-cell adhesion. This study aimed to determine the role of CD44, proliferating cell nuclear antigen (PCNA), and E-cadherin in pterygium formation and recurrence.

DETAILED DESCRIPTION:
Methods:60 patients with pterygium will be enrolled in the study and conjunctival samples will be collected from 30 patients to form the control group. CD44, PCNA and E-cadherin expressions in surgically removed pterygium will be compared with tissue samples from normal control group.

IBM SPSS (statistical software) version 26.0 will be used for statistical analyses.

ELIGIBILITY:
Inclusion Criteria: patient with pterygium -

Exclusion Criteria: patient with pseudopterygium

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 60 patient with primary and recurrent pterygium
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Immunohistochemistry | up to three weeks after pterygium surgery
  Thin sections will be taken from paraffin embedded tissue samples and placed on barcode glass slides After deparaffinization and rehydration, the sections will be subjected to histopathological evaluation using hematoxylin and eosin staining.We use primary antibodies against CD44 (1:50 dilution) and E-cadherin (1:200 dilution), and a human monoclonal antibody against PCNA (1:100 dilution) for antigen retrieval

CONTACTS AND LOCATIONS:
Overall Officials: HÜMEYRA YILDIRIM, Principal Investigator — Balıkesir Medical Faculty
Locations (1):
- Hümeyra Yildirim, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No